CLINICAL TRIAL: NCT05402020
Title: Effectiveness of Maintenance Treatment With Tiotropium + Olodaterol in Comparison to Inhaled Corticosteroids + Long-acting β2 Agonists in COPD Patients in Taiwan: a Non-interventional Study Based on the Taiwan National Health Insurance (NHI) Data
Brief Title: Effectiveness of Tiotropium + Olodaterol Versus Inhaled Corticosteroids (ICS) + Long-acting β2-agonists (LABA) Among COPD Patients in Taiwan
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0110
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tiotropium + Olodaterol cohort: Subjects who initiated Tiotropium + Olodaterol between 1st January 2014 and 31st December 2019 according to data from the Taiwan National Health Insurance (NHI), Taiwan Cancer Registry (TCR) and Taiwan Mortality Data.
  Interventions: Drug: Tiotropium (Tio); Drug: Olodaterol (Olo)
- Inhaled Corticosteroids (ICS) + Long-acting ß2 agonists (LABA) cohort: Subjects who initiated Inhaled Corticosteroids (ICS) + Long-acting ß2 agonists (LABA) between 1st January 2014 and 31st December 2019 according to data from the Taiwan National Health Insurance (NHI), Taiwan Cancer Registry (TCR) and Taiwan Mortality Data.
  Interventions: Drug: Inhaled corticosteroids (ICS); Drug: Long-acting β2-agonists (LABA)

INTERVENTIONS:
Drug: Tiotropium (Tio) — Tiotropium (Tio)
  Groups: Tiotropium + Olodaterol cohort
Drug: Inhaled corticosteroids (ICS) — Inhaled corticosteroids (ICS)
  Groups: Inhaled Corticosteroids (ICS) + Long-acting ß2 agonists (LABA) cohort
Drug: Olodaterol (Olo) — Olodaterol (Olo)
  Groups: Tiotropium + Olodaterol cohort
Drug: Long-acting β2-agonists (LABA) — Long-acting β2-agonists (LABA)
  Groups: Inhaled Corticosteroids (ICS) + Long-acting ß2 agonists (LABA) cohort

SUMMARY:
The real world study aims to assess effectiveness and safety profile between tiotropium/olodaterol (Tio/Olo) and inhaled corticosteroids(ICS) / Long-acting β2-agonists (LABA) in patients with chronic obstructive pulmonary disease (COPD) in Taiwan. The data used in this study will come from the Taiwan National Health Insurance (NHI) claims data between 2014 and 2019.

ELIGIBILITY:
Inclusion Criteria:

1. At least one prescriptions for Tiotropium/Olodaterol (Tio/Olo) combined inhaler or Long-acting ß2 agonist / Inhaled Corticosteroids (LABA/ICS) combined inhaler between 1st January 2014 and 31st December 2019.

   1. The first dispensing of either Tio/Olo or LABA/ICS combined inhaler will be defined as the index date;
   2. For the main analyses, only fixed dose combination (FDC) inhalers will be included.
2. Aged ≥ 40 years on the index date (in a sensitivity analysis we will only include patients aged ≥ 55 years on the index date);
3. At least one diagnosis of chronic obstructive pulmonary disease (COPD) at any time prior to or on the index date;
4. At least one year of continuous medical and health insurance plan prior to the index date will be required to allow for a look-back period for the covariates and identification of new use of the study drugs;
5. At least one record in the health insurance system database

Exclusion Criteria:

1. Any use of Tio/Olo, ICS/LABA, or ICS/LABA/ Long-acting muscarinic antagonists (LAMA) in free or fixed form for one year prior to the index date;
2. Individuals with asthma, allergic rhinitis, lung cancer, interstitial lung disease, or lung transplant identified at any time prior to the index date (in a sensitivity analysis we will include patients with asthma);

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive pulmonary disease, included in the NHI database between 2014 and 2019, who received either Tiotropium + Olodaterol or Inhaled Corticosteroids + Long-acting ß2 agonist.
Sampling Method: Non-Probability Sample
Enrollment: 17018 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Tawain University Hospital, Taipei, China

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/msw/datatransparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a real-world study to assess effectiveness and safety profiles between tiotropium/olodaterol (Tio/Olo) and Inhaled Corticosteroids (ICS) + Long-acting ß2 agonists (LABA). Data sources included Taiwan National Health Insurance (NHI), Taiwan Cancer Registry (TCR) and Taiwan Mortality Data.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated. Only subjects that met all inclusion and none of the exclusion criteria were included in the study.
Period: Overall Study
Arm/Group | Tiotropium + Olodaterol Cohort | Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort
Started | 3815 | 13203
Propensity Score-matched Cohorts | 3752 | 3752
Completed | 3815 | 13203
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Propensity score matched cohorts: Subjects were 1:1 propensity score matched between cohorts. The two groups were comparable with regards to year of treatment initiation, season of treatment initiation, prior treatment for COPD, use of respiratory drugs of interest, frequency and severity of Chronic Obstructive Pulmonary Disease (COPD) exacerbation, prevalence of major comorbidity, Charlson Comorbidity Index, and concomitant medications.
Groups:
- Tiotropium + Olodaterol Cohort - Propensity Score Matched: Subjects who initiated Tiotropium + Olodaterol between 1st January 2014 and 31st December 2019 according to data from the Taiwan National Health Insurance (NHI), Taiwan Cancer Registry (TCR) and Taiwan Mortality Data.
  Subjects were 1:1 propensity score matched to the ICS + LABA cohort. The two groups were comparable with regards to year of treatment initiation, season of treatment initiation, prior treatment for Chronic Obstructive Pulmonary Disease (COPD), use of respiratory drugs of interest, frequency and severity of COPD exacerbation, prevalence of major comorbidity, Charlson Comorbidity Index, and concomitant medications.
- Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched: Subjects who initiated Inhaled Corticosteroids (ICS) + Long-acting ß2 agonists (LABA) between 1st January 2014 and 31st December 2019 according to data from the Taiwan National Health Insurance (NHI), Taiwan Cancer Registry (TCR) and Taiwan Mortality Data.
  Subjects were 1:1 propensity score matched to the Tiotropium + Olodaterol cohort. The two groups were comparable with regards to year of treatment initiation, season of treatment initiation, prior treatment for Chronic Obstructive Pulmonary Disease (COPD), use of respiratory drugs of interest, frequency and severity of COPD exacerbation, prevalence of major comorbidity, Charlson Comorbidity Index, and concomitant medications.
- Total: Total of all reporting groups
Arm/Group | Tiotropium + Olodaterol Cohort - Propensity Score Matched | Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched | Total
Number analyzed (Participants) | 3752 | 3752 | 7504
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (12.19) | 72 (12.76) | 72 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 451 | 458 | 909
  Male | 3301 | 3294 | 6595
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Event First Moderate or Severe COPD Exacerbations After Index Date
Description: Number of subjects with event first moderate or severe COPD exacerbations after index date. The first dispensing of either Tio/Olo or ICS/LABA combined inhaler was defined as the index date.
  Definition of moderate or severe COPD exacerbation:
  1. Moderate exacerbation was defined as an outpatient visit with a diagnosis code for COPD in any field and a prescription for an oral corticosteroid or an antibiotic for respiratory infections
  2. Severe exacerbation was defined as a hospitalization or emergency room visit with a primary diagnosis for COPD
Time Frame: From the index date (the first dispensing of either Tio/Olo or ICS/LABA combined inhaler) until first event, up to 6 years.
Population: Propensity score matched cohorts: Subjects were 1:1 propensity score matched between cohorts. The two groups were comparable with regards to year of treatment initiation, season of treatment initiation, prior treatment for Chronic Obstructive Pulmonary Disease (COPD), use of respiratory drugs of interest, frequency and severity of COPD exacerbation, prevalence of major comorbidity, Charlson Comorbidity Index, and concomitant medications.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium + Olodaterol Cohort - Propensity Score Matched | Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched
Number analyzed (Participants) | 3752 | 3752
Participants | 424 | 375
Statistical Analysis 1: Comparison: Tiotropium + Olodaterol Cohort - Propensity Score Matched vs Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched; Univariate proportional hazards regression was used to compare the time to event (first moderate or severe COPD exacerbations) between the two treatment groups. In the event that there were baseline covariates with unequal distribution between the treatment groups, defined as absolute standardized difference larger than 0.1, the covariate(s) were included in a multiple regression model in addition to the exposure status (Tio/Olo or ICS/LABA); Test type: Other; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.87 to 1.15] — Ratio calculated as [Tio/Olo]/[ICS/LABA]

2. Secondary Outcome: Number of Subjects With Event Triple Therapy Escalation After Index Date
Description: Number of subjects with event triple therapy escalation, defined as any LAMA/ICS/LABA fixed dose combination or any concurrent use for 30 consecutive days of the following:
  1. any LAMA/LABA fixed dose combination + any ICS single formulation
  2. any LAMA single formulation + any ICS/LABA fixed dose combination
  3. any LAMA single formulation + any LABA single formulation + any ICS single formulation
  The event date was the 30th day after initiation of triple therapy.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium + Olodaterol Cohort - Propensity Score Matched | Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched
Number analyzed (Participants) | 3752 | 3752
Participants | 122 | 153
Statistical Analysis 1: Comparison: Tiotropium + Olodaterol Cohort - Propensity Score Matched vs Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched; Univariate proportional hazards regression was used to compare the time to event (triple therapy escalation) between the two treatment groups. In the event that there were baseline covariates with unequal distribution between the treatment groups, defined as absolute standardized difference larger than 0.1, the covariate(s) were included in a multiple regression model in addition to the exposure status (Tio/Olo or ICS/LABA); Test type: Other; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.53 to 0.85] — Ratio calculated as [Tio/Olo]/[ICS/LABA]

3. Secondary Outcome: Incidence Rate of Triple Therapy Initiation
Description: Incidence rate of triple therapy initiation (first event per patient). Triple therapy escalation, defined as any LAMA/ICS/LABA fixed dose combination or any concurrent use for 30 consecutive days of the following:
  1. any LAMA/LABA fixed dose combination + any ICS single formulation
  2. any LAMA single formulation + any ICS/LABA fixed dose combination
  3. any LAMA single formulation + any LABA single formulation + any ICS single formulation
  Incidence rate calculated as (total number of patients in the cohort experiencing an event of interest for the first time during the given time period) / (total person-time at risk from current use of treatment of cohort during the given period).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events(escalations per 1000 person years
Arm/Group | Tiotropium + Olodaterol Cohort - Propensity Score Matched | Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched
Number analyzed (Participants) | 3752 | 3752
Events(escalations per 1000 person years | 76.2 [74.5 to 77.9] | 114.2 [112.1 to 116.3]
Statistical Analysis 1: Comparison: Tiotropium + Olodaterol Cohort - Propensity Score Matched vs Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched; The rate ratio of Tio+Olo - exposed group relative to LABA/ICS group, along with 95% CIs were derived using a univariate negative binomial model. In the event that there are baseline covariates with unequal distribution between the treatment groups, defined as absolute standardized difference larger than 0.1, the covariate(s) will be included in a multiple regression model in addition to the exposure status (Tio/Olo or LABA/ICS); Test type: Other; Incidence difference = -37.9, 95% CI 2-sided [-60.1 to -15.8] — Incidence difference calculated as [incidence rate of Tio/Olo]-[incidence rate of ICS/LABA]
Statistical Analysis 2: Comparison: Tiotropium + Olodaterol Cohort - Propensity Score Matched vs Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched; [analysis description as in outcome 3, analysis 1]; Test type: Other; Incidence Rate Ratio = 0.66, 95% CI 2-sided [0.51 to 0.85] — Ratio calculated as [incidence rate of Tio/Olo]/[incidence rate of ICS/LABA]

4. Secondary Outcome: Number of Subjects With Event First Hospitalization for Community-acquired Pneumonia After Entry
Description: Number of subjects with event the first hospitalization for community-acquired pneumonia after initiation of study drug.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium + Olodaterol Cohort - Propensity Score Matched | Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched
Number analyzed (Participants) | 3752 | 3752
Participants | 11 | 11
Statistical Analysis 1: Comparison: Tiotropium + Olodaterol Cohort - Propensity Score Matched vs Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched; Univariate proportional hazards regression was used to compare the time to event (first hospitalization for community-acquired pneumonia after initiation of study drug) between the two treatment groups. In the event that there were baseline covariates with unequal distribution between the treatment groups, defined as absolute standardized difference larger than 0.1, the covariate(s) were included in a multiple regression model in addition to the exposure status (Tio/Olo or ICS/LABA); Test type: Other; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.36 to 1.93] — Ratio calculated as [Tio/Olo]/[ICS/LABA]

5. Secondary Outcome: Annualized Rate of Prescriptions of Rescue Medications After the Index Date
Description: Annualized rate of prescriptions of rescue medications after the index date. Rescue medications were defined as free or combination use of short-acting beta-agonist (SABA) or short-acting muscarinic antagonist (SAMA) or SABA/SAMA.
  Annualized rates were calculated for each cohort as follows: (total number of events in the cohort during the given time period) / (total person-year at risk from current use of treatment of cohort during the given period).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events (prescriptions) per Person-year
Arm/Group | Tiotropium + Olodaterol Cohort - Propensity Score Matched | Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched
Number analyzed (Participants) | 3752 | 3752
Events (prescriptions) per Person-year | 0.86 [0.01 to 5.33] | 1.03 [0.03 to 5.62]
Statistical Analysis 1: Comparison: Tiotropium + Olodaterol Cohort - Propensity Score Matched vs Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched; [analysis description as in outcome 3, analysis 1]; Test type: Other; Annualized rate ratio = 0.92, 95% CI 2-sided [0.81 to 1.03] — Annualized rate ratio calculated as [annualized rate of Tio/Olo]/[annualized rate of ICS/LABA]

6. Secondary Outcome: Annualized Rate of COPD Exacerbations After Index Date
Description: Annualized rate of moderate or severe COPD exacerbation after the index date. Annualized rate is calculated as follows: number of moderate or severe COPD exacerbations/total patient year at risk=number of exacerbations per patient year.
  Definitions of moderate or severe COPD exacerbation were:
  1. Moderate exacerbation was defined as an outpatient visit with a diagnosis code for COPD in any field + a prescription for an oral corticosteroid or an antibiotic for respiratory infections, prescriptions within 30 days of each other were considered as continuation of the initial exacerbation.
  2. Severe exacerbation was defined as a hospitalization or emergency room visit with a primary diagnosis for COPD; hospitalizations or emergency room visits within 30 days of each other were considered as continuation of the initial exacerbation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events (exacerbations) per Person-year
Arm/Group | Tiotropium + Olodaterol Cohort - Propensity Score Matched | Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched
Number analyzed (Participants) | 3752 | 3752
Events (exacerbations) per Person-year | 0.36 [0.00 to 4.41] | 0.37 [0.00 to 4.42]
Statistical Analysis 1: Comparison: Tiotropium + Olodaterol Cohort - Propensity Score Matched vs Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort - Propensity Score Matched; [analysis description as in outcome 3, analysis 1]; Test type: Other; Annualized rate ratio = 1.01, 95% CI 2-sided [0.87 to 1.18] — Annualized rate ratio calculated as [annualized rate of Tio/Olo]/[annualized rate of ICS/LABA]

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study.
Description: This is a non-interventional study using electronic health care records, with data retrieved from Danish National Patient Registry, Danish National Prescription Registry and Danish Register of Causes of Death. No adverse events were collected on an individual case level.
Arm/Group | Tiotropium + Olodaterol Cohort | Inhaled Corticosteroids (ICS) + Long-acting ß2 Agonists (LABA) Cohort
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Clinically important parameters and reasons for using medications were not available. Anticipated is that a certain level of misclassification of disease conditions occurred. Not accounting for such confounders may have resulted in biased findings. Follow-up was censored resulting in limited follow-up time. This may have compromised statistical power, but was not likely to contribute substantial bias in the comparisons. SEAP template does not contain a document date as per internal SOP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT05402020/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT05402020/SAP_001.pdf